CLINICAL TRIAL: NCT07230847
Title: A Study Evaluating the Vascular Healing and Neointimal Transformation at 1 Month After Implantation of BioFreedom™ Drug-coated Stents and the Xience Drug-eluting Stent System in Patients With Acute Coronary Syndrome and High Bleeding Risk Using Optical Coherence Tomography
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-ZX094
Record Dates: First submitted 2025-09-28; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-09

CONDITIONS: Coronary Heart Disease; Acute Coronary Syndrome
MeSH Terms: conditions — Coronary Disease; Acute Coronary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BioFreedom™ Drug-Coated Coronary Stent Intervention Group (Experimental)
  Interventions: Device: BioFreedom™
- Xience Drug-Eluting Coronary Stent System Intervention Group (Active Comparator)
  Interventions: Device: Xience

INTERVENTIONS:
Device: BioFreedom™ — BioFreedom™ Drug-Coated Coronary Stent Intervention
  Arms: BioFreedom™ Drug-Coated Coronary Stent Intervention Group
Device: Xience — Xience Drug-Eluting Coronary Stent System Intervention
  Arms: Xience Drug-Eluting Coronary Stent System Intervention Group

SUMMARY:
BioFreedom™ is the world's first polymer-free drug-coated stent (DCS), utilizing a proprietary microstructured surface technology. Its abluminal microporous surface directly carries BA9™ (a sirolimus derivative) with high lipophilicity. This design mitigates inflammatory responses while promoting early vascular healing and reducing thrombotic risk. Extensive clinical evidence has validated BioFreedom™'s superior performance in high-bleeding-risk (HBR) populations. However, comprehensive assessments of neointimal coverage and quantitative neointimal transformation post-implantation remain insufficient. With advancements in ultra-high-resolution optical coherence tomography (OCT), detailed evaluation of coronary stent healing has become feasible. This study will employ OCT to comparatively assess vascular healing patterns-including neointimal transformation and strut coverage-in ACS patients with HBR receiving either the commercially available BioFreedom™ DCS or Xience drug-eluting stent system. The findings will provide multidimensional insights into the devices' post-implantation efficacy and safety profiles.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Male or non-pregnant female
3. Acute coronary syndrome (ACS) patients requiring percutaneous coronary intervention (PCI)
4. No contraindications for coronary artery bypass grafting (CABG)
5. High bleeding risk (HBR) patients per ARC-HBR definition (meeting ≥1 major or 2 minor criteria):

   Major Criteria:
   * Expected long-term oral anticoagulation
   * Severe/end-stage chronic kidney disease (eGFR <30 mL/min)
   * Moderate/severe anemia (Hb <110 g/L)
   * Spontaneous bleeding requiring hospitalization/transfusion within 6 months (or recurrent)
   * Chronic bleeding diathesis
   * Moderate/severe thrombocytopenia pre-PCI (platelet count <100×10⁹/L)
   * Liver cirrhosis with portal hypertension
   * Active malignancy in past 12 months (excluding non-melanoma skin cancer; defined as diagnosis/treatment within 12 months)
   * History of spontaneous intracranial hemorrhage
   * Traumatic intracranial hemorrhage within 12 months
   * Known cerebral arteriovenous malformation
   * Moderate/severe ischemic stroke within 6 months
   * Major surgery/severe trauma within 30 days pre-PCI
   * Planned non-deferrable major surgery during dual antiplatelet therapy

   Minor Criteria:
   * Age ≥75 years
   * Moderate chronic kidney disease (eGFR:30~59 ml/min)
   * Mild anemia (male: Hb=110~129 g/L; female: Hb=110~119 g/L)
   * Spontaneous bleeding requiring hospitalization/transfusion within 6-12 months pre-PCI
   * Chronic NSAID/steroid use post-PCI
   * Ischemic stroke >6 months pre-PCI
6. Capable of understanding trial objectives and providing informed consent

Angiographic Inclusion Criteria:

1. Target lesion must be primary native coronary artery lesion
2. Target lesion with ≥70% diameter stenosis (visual estimate), or 50-70% diameter stenosis (visual estimate) with ischemic evidence
3. ≥1 non-target lesion requiring intervention
4. Non-target lesions eligible for elective treatment within 1 month

Exclusion Criteria:

General Exclusion Criteria:

1. Presence of ≥1 evidence of heart failure including:

   * NYHA Class III or higher, or
   * Killip classification ≥ Grade 2, or
   * Left ventricular ejection fraction (LVEF) ≤30% within 30 days pre-procedure (by echocardiography or intraoperative ventriculography)
2. Cardiogenic shock patients
3. Known allergies to: Aspirin / clopidogrel / ticagrelor / heparin, Contrast agents/drugs used in drug-eluting stents or contraindications to aspirin/ clopidogrel / ticagrelor
4. Life expectancy <12 months or factors potentially compromising clinical follow-up
5. Participation in other drug/medical device trials prior to enrollment without reaching primary endpoint timelines
6. History of substance abuse (alcohol/cocaine/heroin, etc.)
7. Severe arrhythmias (e.g., high-risk ventricular premature contractions/ ventricular tachycardia)
8. Other medical conditions deemed unsuitable by investigators

Angiographic Exclusion Criteria:

1. Left main coronary artery disease
2. Bypass graft lesions
3. Evidence of extensive thrombus in target vessel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
OCT-Detected Neointimal Strut Coverage at 1-Month Post-Procedure | 1-Month Post-Procedural Follow-Up
  Neointimal strut coverage was defined as:
  Covered strut proportion =Number of struts covered by neointima / Total number of analyzable struts A strut is considered covered when both its luminal surface and lateral sides demonstrate continuous neointimal tissue encapsulation.

SECONDARY OUTCOMES:
Neointimal thickness at 1-month post-procedure | 1-Month Post-Procedural Follow-Up
  Strut neointimal thickness (NIT) will be analysed every 1 mm at 1-month post-procedure OCT follow-up
Neointimal area at 1-month post-procedure | 1-Month Post-Procedure Follow-Up
  Lumen area and stent area will be analysed every 1 mm at 1-month post-procedure OCT follow-up, neointimal area (NIA) will be calculated as stent minus lumen area.
Neointimal volume at 1-month post-procedure | 1-Month Post-Procedure Follow-Up
  Neointimal volume (NIV) and stent volume will be calculated using Simpson's rule and reported as total NIV, mean NIV (total NIV divided by length), and percent NIV (NIV divided by stent volume)
Incidence of Major Adverse Cardiac Events (MACE) within 12 Months Post-Procedure | 12 Months Post-Procedure
  MACE is defined as a composite of cardiac death, myocardial infarction, and target vessel revascularization (TVR).
Incidence of stent thrombosis within 12 months post-procedure | 12 Months Post-Procedure
  Stent thrombosis refers to definite or probable stent thrombosis as defined by the Academic Research Consortium (ARC) criteria
Incidence of bleeding events within 12 months post-procedure | 12 Months Post-Procedure
  bleeding events including BARC types 2, 3, or 5 bleeding.

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai hospital, CAMS&PUMC, Beijing, Beijing Municipality, China